CLINICAL TRIAL: NCT04552366
Title: A Clinical Trial to Evaluate the Safety and Immunogenicity of a Recombinant Adenovirus 5 Vectored COVID-19 Vaccine (Ad5-nCoV) With Two Doses in Healthy Adults Aged 18 Years and Older
Brief Title: A Clinical Trial of a Recombinant Adenovirus 5 Vectored COVID-19 Vaccine (Ad5-nCoV) With Two Doses in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Biotechnology, Academy of Military Medical Sciences, PLA of China (Other)
Collaborators: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AMMS85-2004
Record Dates: First submitted 2020-09-15; First posted 2020-09-17 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: COVID-19
Keywords: COVID-19 vaccine; Ad5-nCoV
MeSH Terms: conditions — COVID-19 | interventions — Ad5-nCoV vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group A: Intramuscular administration (Experimental): 24 subjects. 5E10 VP of Ad5-nCoV on Day 0 and on Day 56.
  Interventions: Biological: Ad5-nCoV
- Group B: Mixed administration (Experimental): 24 subjects. An intramuscular administration of 5E10 VP of Ad5-nCoV on day 0 and a mucosal administration of 2E10 VP on Day 28.
  Interventions: Biological: Ad5-nCoV
- Group C: Mucosal administration, high dose (Experimental): 24 subjects. A mucosal administration of 2E10 VP of Ad5-nCoV on Day 0 and Day 28.
  Interventions: Biological: Ad5-nCoV
- Group D: Mucosal administration, low dose (Experimental): 24 subjects. A mucosal administration of 1E10 VP of Ad5-nCoV on day 0 and Day 28.
  Interventions: Biological: Ad5-nCoV
- Group E: Intramuscular administration, one dose (Active Comparator): 24 subjects. An intramuscular administration of 5E10 VP of Ad5-nCoV on day 0.
  Interventions: Biological: Ad5-nCoV
- Group F: Intramuscular administration, two doses (Experimental): 24 subjects. Two intramuscular administrations of 5E10 VP of Ad5-nCoV at left and right arms on day 0.
  Interventions: Biological: Ad5-nCoV

INTERVENTIONS:
Biological: Ad5-nCoV — Recombinant Novel Coronavirus Vaccine (Adenovirus Type 5 Vector)

SUMMARY:
This is a clinical trial to evaluate the safety and immunogenicity of a recombinant adenovirus 5 vectored COVID-19 vaccine (Ad5-nCoV) with two doses and with different adminstration routes in healthy adults aged 18 years and older.

DETAILED DESCRIPTION:
A total of 168 healthy adult volunteers will be vaccinated in this clinical trial according to open, partly randomized design from the healthy adults aged 18 years and older. The safety and immunogenicity of intramuscular vaccination and mucosal vaccination of two doses of Ad5-nCoV in different administration schedules will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years and older;
* Able to provide consent to participate in and having signed an Informed Consent Form (ICF);
* Able and willing to complete all the scheduled study procedures during the whole study follow-up period (about 6-8 months, depending on group);
* Negative result of HIV screening;
* Axillary temperature ≤37.0°C.
* Negative IgG and IgM antibodies against COVID-19;
* Good general health status, as determined by history and physical examination.

Exclusion Criteria for the first vaccination:

* Hematological examination is abnormal, or clinically significant as assessed by the study investigator (including white blood cell count, lymphocyte count, neutrophil count, eosinophil count, platelet, hemoglobin, alanine aminotransferase (ALT), aspartate aminotransferase (AST), total bilirubin, blood glucose and creatinine);
* With oral ulcers, throat swelling and other oral diseases.
* With symptoms of upper respiratory tract infection.
* Personal history of seizure disorder, encephalopathy or psychosis;
* Allergic history to any vaccine, or allergic to any ingredient of the Ad5-nCoV;
* Any acute febrile disease or active infectious disease on the day of vaccination;
* History of SARS or COVID-19;
* History of COVID-19 candidate vaccine administration;
* History of chronic obstructive pulmonary disease (COPD).
* Serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, severe hypertension not controlled with medication;
* Serious chronic disease or in the advanced stage that cannot be controlled well， such as asthma, diabetes and thyroid disease, etc.;
* Congenital or acquired angioedema;
* Suffered from urticaria within 1 year before receiving the trial vaccine.
* Asplenia or functional asplenia;
* Platelet disorder or other bleeding disorder that may cause intramuscular injection contraindication;
* Faint with needles in intramuscular administration group;
* Immunosuppressive medication, anti-allergic, cytotoxic therapy, inhaled corticosteroids (excluding surface corticosteroid therapy for acute non-complicated dermatitis) in the last 6 months;
* Prior administration of blood products in last 4 months;
* Other vaccination(s) or investigational drugs within 1 month before study onset;
* Prior administration of live attenuated vaccine within 1 month before study onset;
* Prior administration of subunit or inactivated vaccine within 14 days before study onset;
* Current anti-tuberculosis therapy;
* Woman is pregnant or lactating, positive urine pregnancy test or plan to become pregnant during the next 8 months;
* Any condition that in the opinion of the investigators may interfere with the participants' compliance or evaluation of study objectives or informed consent (i.e. medical, psychological, social or other conditions, etc.).

Exclusion Criteria for the second vaccination:

* Severe allergic reaction after the first dose of vaccination;
* Severe adverse reactions causally related to the first vaccination;
* For those newly discovered or newly occured after the first vaccination that does not meet the first-dose selection criteria or meets the first-dose exclusion criteria, the investigator will determine whether to continue participating in the study;
* Other reasons for exclusion as deemed by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Incidence of the AE in all groups | 0-7 days after each vaccination
  The occurrence of AE in all groups within 0-7 days after each vaccination;
Seroconversion rate of the IgG antibody against SARS-CoV-2 | Day 28 after last vaccination
  Seroconversion rate the IgG antibody against SARS-CoV-2 measured on Day 28 after last vaccination
Geomean titers of the IgG antibody against SARS-CoV-2 | Day 28 after last vaccination
  Geomean titers of the IgG antibody against SARS-CoV-2 measured on Day 28 after last vaccination
Seroconversion rate of the neutralizing antibody against SARS-CoV-2 | Day 28 after last vaccination
  Seroconversion rate of the neutralizing antibody against SARS-CoV-2 measured on Day 28 after last vaccination
Geomean titers of the neutralizing antibody against SARS-CoV-2 | Day 28 after last vaccination
  Geomean titers of the neutralizing antibody against SARS-CoV-2 measured on Day 28 after last vaccination

SECONDARY OUTCOMES:
Incidence of the AE in all groups | 0-30 minutes, 0-28 days after each vaccination
  The occurrence of AE in all groups within 0-30 minutes and 0-28 days after each vaccination.
Incidence of Serious adverse events (SAE) in all groups | 6 months after the final vaccination
  The occurrence of Serious adverse events (SAE) in all groups within 6 months after the final vaccination.
Geomean titers of the IgG antibody against SARS-CoV-2 | Day 0, 14, 28 and 56 after first vaccination and Day 14 and Day168 after last vaccination.
  Geomean titers of the IgG antibody against SARS-CoV-2 measured on Day 0, 14, 28 and 56 after first vaccination and on Day 14 and Day168 after last vaccination.
Seroconversion rate of the IgG antibody against SARS-CoV-2 | Day 0, 14, 28 and 56 after first vaccination and Day 14 and Day168 after last vaccination.
  Seroconversion rate of the IgG antibody against SARS-CoV-2 measured on Day 0, 14, 28 and 56 after first vaccination and on Day 14 and Day168 after last vaccination.
Geomean titers of the neutralizing antibody against SARS-CoV-2 | Day 0, 14, 28 and 56 after first vaccination and Day 14 and Day168 after last vaccination.
  Geomean titers of the neutralizing antibody against SARS-CoV-2 measured on Day 0, 14, 28 and 56 after first vaccination and on Day 14 and Day168 after last vaccination.
Seroconversion rate of the neutralizing antibody against SARS-CoV-2 | Day 0, 14, 28 and 56 after first vaccination and on Day 14 and Day168 after last vaccination.
  Seroconversion rate of the neutralizing antibody against SARS-CoV-2 measured on Day 0, Day14, Day 28 or Day 56 after first vaccination and on day 14, day 28 and day168 after last vaccination.
Cellular immune response by ELISpot | Day 0 and Day 14 after each vaccination
  The positive rate of IFN-γ stimulated by S protein overlapping peptide library detected by ELISpot on Day 0 and Day 14 after each vaccination
Geomean titers of neutralizing antibody response to Ad5-vector | Day 0, 14 and 28 after each vaccination.
  Geomean titers of neutralizing antibody response to Ad5-vector on Day 0, 14 and 28 after each vaccination.
Cellular immune response by ICS | Day 0 and Day 14 after each vaccination
  The positive rate of the specific cytokines expressed by CD4+ and CD8+ T lymphocytes stimulated by S protein overlapping peptide library detected by intracellular cytokine staining on Day 0 and Day 14 after each vaccination
Geomean titers of the IgA antibody against SARS-CoV-2 | Day 0, 14 and 28 after each vaccination
  Geomean titers of the IgA antibody against SARS-CoV-2 on Day 0, 14 and 28 after each vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongnan Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu S, Huang J, Zhang Z, Wu J, Zhang J, Hu H, Zhu T, Zhang J, Luo L, Fan P, Wang B, Chen C, Chen Y, Song X, Wang Y, Si W, Sun T, Wang X, Hou L, Chen W. Safety, tolerability, and immunogenicity of an aerosolised adenovirus type-5 vector-based COVID-19 vaccine (Ad5-nCoV) in adults: preliminary report of an open-label and randomised phase 1 clinical trial. Lancet Infect Dis. 2021 Dec;21(12):1654-1664. doi: 10.1016/S1473-3099(21)00396-0. Epub 2021 Jul 26. PMID 34324836